CLINICAL TRIAL: NCT01413009
Title: Awakening-Breathing Coordination, Delirium Monitoring/Management & Early Mobility (ABCDE) Protocol
Acronym: ABCDE
Status: Completed | Type: Observational
Sponsor: University of Nebraska (Other)
Collaborators: Robert Wood Johnson Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 0590-10-FB
Record Dates: First submitted 2011-08-02; First posted 2011-08-09 (Estimated); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: ICU Delirium; Immobility
Keywords: delirium; ICU; spontaneous awakening trials; spontaneous breathing trials; early mobility
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ICU patients: Adult patients admitted to the University of Nebraska Medical Center or the Nebraska Medical Center trauma critical care service.

SUMMARY:
Fully two-thirds of ICU patients develop delirium, which is associated with longer stays, billions of dollars in costs globally, and 3-fold excess mortality at 6 months. Over one-half of ICU survivors suffer a functionally debilitating dementia-like illness, which appears related to delirium duration. This study will focus on applying Awakening-Breathing Coordination, Delirium Monitoring/Management & Early Mobility (ABCDE), a program of delirium screening, prevention, and treatment developed at Vanderbilt University. Specifically, the study will implement the ABCDE program in a medical center that does not currently perform routine ICU delirium screenings and identify facilitators and barriers to program adoption; test the impact of the ABCDE program on patient outcomes, nursing quality outcomes, and system outcomes; and assess the extent to which ABCDE implementation is effective, sustainable, and conducive to dissemination into other settings.

DETAILED DESCRIPTION:
We face a profound and emerging public health problem in the form of acute and chronic brain dysfunction among young and elderly intensive care unit (ICU) survivors that is altering the landscape of society. Fully two-thirds of ICU patients develop delirium, which is associated with longer stays, billions of dollars in costs globally, and 3-fold excess mortality at 6 months. Over one-half of ICU survivors suffer a functionally debilitating dementia-like illness, which appears related to delirium duration. The impact on a person's life is often devastating. The main goal of the proposed INQRI project is to implement, analyze, and disseminate an evidence-based, nurse-led, inter-professional, multi-component program focused on improving the care and outcomes of critically ill adults. The study will focus on applying Awakening-Breathing Coordination, Delirium Monitoring/Management & Early Mobility (ABCDE), a program of delirium screening, prevention, and treatment developed at Vanderbilt University. The ABCDE approach analyzes and merges the best available evidence related to delirium, analgesia, and sedation (DAS) management in the ICU and tailors the pharmacologic and nonpharmacologic interventions used in prior DAS clinical trials into a program that can be adopted into practice in less "research focused" ICUs. Specifically, the study aims are to (1) implement the ABCDE program in a medical center that does not currently perform routine ICU delirium screenings and identify facilitators and barriers to program adoption; (2) test the impact of the ABCDE program on patient outcomes, nursing quality outcomes, and system outcomes; and (3) assess the extent to which ABCDE implementation is effective, sustainable, and conducive to dissemination into other settings.

ELIGIBILITY:
Inclusion Criteria:

* Greater than or equal to 19 years of age
* Patients at the University of Nebraska Medical Center and the Nebraska Medical Center
* Admitted to either the academic medical or trauma critical care service

Exclusion Criteria:

* Legally authorized representative not available to provide consent to participate within 48 hours of ICU admission

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critical care services
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2010-12-29 (Actual); Primary Completion 2012-04-01 (Actual); Study Completion 2013-06-01 (Actual)

PRIMARY OUTCOMES:
Ventilator free days (VFDs) | Change in ventlator free days at baseline to 9 months
  The primary outcome will be a comparison between the 3 month baseline period of ventilator free days and the 9 month period following the intervention. Two interim analyses will be conducted.

CONTACTS AND LOCATIONS:
Overall Officials: Michele Balas, PhD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

REFERENCES:
- [Background] Ely EW, Shintani A, Truman B, Speroff T, Gordon SM, Harrell FE Jr, Inouye SK, Bernard GR, Dittus RS. Delirium as a predictor of mortality in mechanically ventilated patients in the intensive care unit. JAMA. 2004 Apr 14;291(14):1753-62. doi: 10.1001/jama.291.14.1753. PMID 15082703
- [Background] Ely EW, Inouye SK, Bernard GR, Gordon S, Francis J, May L, Truman B, Speroff T, Gautam S, Margolin R, Hart RP, Dittus R. Delirium in mechanically ventilated patients: validity and reliability of the confusion assessment method for the intensive care unit (CAM-ICU). JAMA. 2001 Dec 5;286(21):2703-10. doi: 10.1001/jama.286.21.2703. PMID 11730446
- [Background] Pandharipande P, Cotton BA, Shintani A, Thompson J, Pun BT, Morris JA Jr, Dittus R, Ely EW. Prevalence and risk factors for development of delirium in surgical and trauma intensive care unit patients. J Trauma. 2008 Jul;65(1):34-41. doi: 10.1097/TA.0b013e31814b2c4d. PMID 18580517
- [Background] Lat I, McMillian W, Taylor S, Janzen JM, Papadopoulos S, Korth L, Ehtisham A, Nold J, Agarwal S, Azocar R, Burke P. The impact of delirium on clinical outcomes in mechanically ventilated surgical and trauma patients. Crit Care Med. 2009 Jun;37(6):1898-905. doi: 10.1097/CCM.0b013e31819ffe38. PMID 19384221
- [Background] Milbrandt EB, Deppen S, Harrison PL, Shintani AK, Speroff T, Stiles RA, Truman B, Bernard GR, Dittus RS, Ely EW. Costs associated with delirium in mechanically ventilated patients. Crit Care Med. 2004 Apr;32(4):955-62. doi: 10.1097/01.ccm.0000119429.16055.92. PMID 15071384
- [Background] Sleiman I, Rozzini R, Trabucchi M. Delirium in older patients in intensive care units. Arch Intern Med. 2008 Jun 9;168(11):1229. doi: 10.1001/archinte.168.11.1229-a. No abstract available. PMID 18541836
- [Background] Ouimet S, Kavanagh BP, Gottfried SB, Skrobik Y. Incidence, risk factors and consequences of ICU delirium. Intensive Care Med. 2007 Jan;33(1):66-73. doi: 10.1007/s00134-006-0399-8. Epub 2006 Nov 11. PMID 17102966
- [Background] Thomason JW, Shintani A, Peterson JF, Pun BT, Jackson JC, Ely EW. Intensive care unit delirium is an independent predictor of longer hospital stay: a prospective analysis of 261 non-ventilated patients. Crit Care. 2005 Aug;9(4):R375-81. doi: 10.1186/cc3729. Epub 2005 Jun 1. PMID 16137350
- [Background] Ely EW, Gautam S, Margolin R, Francis J, May L, Speroff T, Truman B, Dittus R, Bernard R, Inouye SK. The impact of delirium in the intensive care unit on hospital length of stay. Intensive Care Med. 2001 Dec;27(12):1892-900. doi: 10.1007/s00134-001-1132-2. Epub 2001 Nov 8. PMID 11797025
- [Background] Micek ST, Anand NJ, Laible BR, Shannon WD, Kollef MH. Delirium as detected by the CAM-ICU predicts restraint use among mechanically ventilated medical patients. Crit Care Med. 2005 Jun;33(6):1260-5. doi: 10.1097/01.ccm.0000164540.58515.bf. PMID 15942341
- [Background] Dubois MJ, Bergeron N, Dumont M, Dial S, Skrobik Y. Delirium in an intensive care unit: a study of risk factors. Intensive Care Med. 2001 Aug;27(8):1297-304. doi: 10.1007/s001340101017. PMID 11511942
- [Background] Balas MC, Happ MB, Yang W, Chelluri L, Richmond T. Outcomes Associated With Delirium in Older Patients in Surgical ICUs. Chest. 2009 Jan;135(1):18-25. doi: 10.1378/chest.08-1456. Epub 2008 Nov 18. PMID 19017895
- [Background] Lin SM, Liu CY, Wang CH, Lin HC, Huang CD, Huang PY, Fang YF, Shieh MH, Kuo HP. The impact of delirium on the survival of mechanically ventilated patients. Crit Care Med. 2004 Nov;32(11):2254-9. doi: 10.1097/01.ccm.0000145587.16421.bb. PMID 15640638
- [Background] Pisani MA, Kong SY, Kasl SV, Murphy TE, Araujo KL, Van Ness PH. Days of delirium are associated with 1-year mortality in an older intensive care unit population. Am J Respir Crit Care Med. 2009 Dec 1;180(11):1092-7. doi: 10.1164/rccm.200904-0537OC. Epub 2009 Sep 10. PMID 19745202
- [Background] Jackson JC, Gordon SM, Hart RP, Hopkins RO, Ely EW. The association between delirium and cognitive decline: a review of the empirical literature. Neuropsychol Rev. 2004 Jun;14(2):87-98. doi: 10.1023/b:nerv.0000028080.39602.17. PMID 15264710
- [Background] Halpern NA, Pastores SM. Critical care medicine in the United States 2000-2005: an analysis of bed numbers, occupancy rates, payer mix, and costs. Crit Care Med. 2010 Jan;38(1):65-71. doi: 10.1097/CCM.0b013e3181b090d0. PMID 19730257
- [Background] Happ MB, Tate J, Garret K. Nursing counts. Focus on: nonspeaking older adults in the ICU: communication will require special strategies. American Journal of Nursing 106(5):29, 2006.
- [Background] Happ MB. Interpretation of nonvocal behavior and the meaning of voicelessness in critical care. Soc Sci Med. 2000 May;50(9):1247-55. doi: 10.1016/s0277-9536(99)00367-6. PMID 10728845
- [Background] Happ MB. Communicating with mechanically ventilated patients: state of the science. AACN Clin Issues. 2001 May;12(2):247-58. doi: 10.1097/00044067-200105000-00008. PMID 11759552
- [Background] Inouye SK, Viscoli CM, Horwitz RI, Hurst LD, Tinetti ME. A predictive model for delirium in hospitalized elderly medical patients based on admission characteristics. Ann Intern Med. 1993 Sep 15;119(6):474-81. doi: 10.7326/0003-4819-119-6-199309150-00005. PMID 8357112
- [Background] Patel RP, Gambrell M, Speroff T, Scott TA, Pun BT, Okahashi J, Strength C, Pandharipande P, Girard TD, Burgess H, Dittus RS, Bernard GR, Ely EW. Delirium and sedation in the intensive care unit: survey of behaviors and attitudes of 1384 healthcare professionals. Crit Care Med. 2009 Mar;37(3):825-32. doi: 10.1097/CCM.0b013e31819b8608. PMID 19237884
- [Background] Pun BT, Ely EW. The importance of diagnosing and managing ICU delirium. Chest. 2007 Aug;132(2):624-36. doi: 10.1378/chest.06-1795. PMID 17699134
- [Background] Girard TD, Pandharipande PP, Ely EW. Delirium in the intensive care unit. Crit Care. 2008;12 Suppl 3(Suppl 3):S3. doi: 10.1186/cc6149. Epub 2008 May 14. PMID 18495054
- [Background] Brook AD, Ahrens TS, Schaiff R, Prentice D, Sherman G, Shannon W, Kollef MH. Effect of a nursing-implemented sedation protocol on the duration of mechanical ventilation. Crit Care Med. 1999 Dec;27(12):2609-15. doi: 10.1097/00003246-199912000-00001. PMID 10628598
- [Background] Richman PS, Baram D, Varela M, Glass PS. Sedation during mechanical ventilation: a trial of benzodiazepine and opiate in combination. Crit Care Med. 2006 May;34(5):1395-401. doi: 10.1097/01.CCM.0000215454.50964.F8. PMID 16540957
- [Background] Chanques G, Jaber S, Barbotte E, Violet S, Sebbane M, Perrigault PF, Mann C, Lefrant JY, Eledjam JJ. Impact of systematic evaluation of pain and agitation in an intensive care unit. Crit Care Med. 2006 Jun;34(6):1691-9. doi: 10.1097/01.CCM.0000218416.62457.56. PMID 16625136
- [Background] Mascia MF, Koch M, Medicis JJ. Pharmacoeconomic impact of rational use guidelines on the provision of analgesia, sedation, and neuromuscular blockade in critical care. Crit Care Med. 2000 Jul;28(7):2300-6. doi: 10.1097/00003246-200007000-00019. PMID 10921556
- [Background] Arias-Rivera S, Sanchez-Sanchez Mdel M, Santos-Diaz R, Gallardo-Murillo J, Sanchez-Izquierdo R, Frutos-Vivar F, Ferguson ND, Esteban A. Effect of a nursing-implemented sedation protocol on weaning outcome. Crit Care Med. 2008 Jul;36(7):2054-60. doi: 10.1097/CCM.0b013e31817bfd60. PMID 18552689
- [Background] Quenot JP, Ladoire S, Devoucoux F, Doise JM, Cailliod R, Cunin N, Aube H, Blettery B, Charles PE. Effect of a nurse-implemented sedation protocol on the incidence of ventilator-associated pneumonia. Crit Care Med. 2007 Sep;35(9):2031-6. doi: 10.1097/01.ccm.0000282733.83089.4d. PMID 17855817
- [Background] Kress JP, Pohlman AS, O'Connor MF, Hall JB. Daily interruption of sedative infusions in critically ill patients undergoing mechanical ventilation. N Engl J Med. 2000 May 18;342(20):1471-7. doi: 10.1056/NEJM200005183422002. PMID 10816184
- [Background] Schweickert WD, Gehlbach BK, Pohlman AS, Hall JB, Kress JP. Daily interruption of sedative infusions and complications of critical illness in mechanically ventilated patients. Crit Care Med. 2004 Jun;32(6):1272-6. doi: 10.1097/01.ccm.0000127263.54807.79. PMID 15187505
- [Background] Girard TD, Kress JP, Fuchs BD, Thomason JW, Schweickert WD, Pun BT, Taichman DB, Dunn JG, Pohlman AS, Kinniry PA, Jackson JC, Canonico AE, Light RW, Shintani AK, Thompson JL, Gordon SM, Hall JB, Dittus RS, Bernard GR, Ely EW. Efficacy and safety of a paired sedation and ventilator weaning protocol for mechanically ventilated patients in intensive care (Awakening and Breathing Controlled trial): a randomised controlled trial. Lancet. 2008 Jan 12;371(9607):126-34. doi: 10.1016/S0140-6736(08)60105-1. PMID 18191684
- [Background] Kress JP, Gehlbach B, Lacy M, Pliskin N, Pohlman AS, Hall JB. The long-term psychological effects of daily sedative interruption on critically ill patients. Am J Respir Crit Care Med. 2003 Dec 15;168(12):1457-61. doi: 10.1164/rccm.200303-455OC. Epub 2003 Oct 2. PMID 14525802
- [Background] King MS, Render ML, Ely EW, Watson PL. Liberation and animation: strategies to minimize brain dysfunction in critically ill patients. Semin Respir Crit Care Med. 2010 Feb;31(1):87-96. doi: 10.1055/s-0029-1246284. Epub 2010 Jan 25. PMID 20101551
- [Background] Jacobi J, Fraser GL, Coursin DB, Riker RR, Fontaine D, Wittbrodt ET, Chalfin DB, Masica MF, Bjerke HS, Coplin WM, Crippen DW, Fuchs BD, Kelleher RM, Marik PE, Nasraway SA Jr, Murray MJ, Peruzzi WT, Lumb PD; Task Force of the American College of Critical Care Medicine (ACCM) of the Society of Critical Care Medicine (SCCM), American Society of Health-System Pharmacists (ASHP), American College of Chest Physicians. Clinical practice guidelines for the sustained use of sedatives and analgesics in the critically ill adult. Crit Care Med. 2002 Jan;30(1):119-41. doi: 10.1097/00003246-200201000-00020. No abstract available. PMID 11902253
- [Background] Kress JP, Pohlman AS, Hall JB. Sedation and analgesia in the intensive care unit. Am J Respir Crit Care Med. 2002 Oct 15;166(8):1024-8. doi: 10.1164/rccm.200204-270CC. No abstract available. PMID 12379543
- [Background] Sessler CN, Pedram S. Protocolized and target-based sedation and analgesia in the ICU. Crit Care Clin. 2009 Jul;25(3):489-513, viii. doi: 10.1016/j.ccc.2009.03.001. PMID 19576526
- [Background] Franck LS, Naughton I, Winter I. Opioid and benzodiazepine withdrawal symptoms in paediatric intensive care patients. Intensive Crit Care Nurs. 2004 Dec;20(6):344-51. doi: 10.1016/j.iccn.2004.07.008. PMID 15567675
- [Background] Shintani AK, Girard TD, Ely EW. Immortal time bias in critical care. Crit Care Med. 2010 Apr;38(4):1229. doi: 10.1097/CCM.0b013e3181ce473d. No abstract available. PMID 20335718
- [Background] Robinson BR, Mueller EW, Henson K, Branson RD, Barsoum S, Tsuei BJ. An analgesia-delirium-sedation protocol for critically ill trauma patients reduces ventilator days and hospital length of stay. J Trauma. 2008 Sep;65(3):517-26. doi: 10.1097/TA.0b013e318181b8f6. PMID 18784563
- [Background] Hooper MH, Girard TD. Sedation and weaning from mechanical ventilation: linking spontaneous awakening trials and spontaneous breathing trials to improve patient outcomes. Crit Care Clin. 2009 Jul;25(3):515-25, viii. doi: 10.1016/j.ccc.2009.04.002. PMID 19576527
- [Background] Esteban A, Alia I, Gordo F, Fernandez R, Solsona JF, Vallverdu I, Macias S, Allegue JM, Blanco J, Carriedo D, Leon M, de la Cal MA, Taboada F, Gonzalez de Velasco J, Palazon E, Carrizosa F, Tomas R, Suarez J, Goldwasser RS. Extubation outcome after spontaneous breathing trials with T-tube or pressure support ventilation. The Spanish Lung Failure Collaborative Group. Am J Respir Crit Care Med. 1997 Aug;156(2 Pt 1):459-65. doi: 10.1164/ajrccm.156.2.9610109. PMID 9279224
- [Background] Ely EW, Baker AM, Dunagan DP, Burke HL, Smith AC, Kelly PT, Johnson MM, Browder RW, Bowton DL, Haponik EF. Effect on the duration of mechanical ventilation of identifying patients capable of breathing spontaneously. N Engl J Med. 1996 Dec 19;335(25):1864-9. doi: 10.1056/NEJM199612193352502. PMID 8948561
- [Background] Jackson JC, Girard TD, Gordon SM, Thompson JL, Shintani AK, Thomason JW, Pun BT, Canonico AE, Dunn JG, Bernard GR, Dittus RS, Ely EW. Long-term cognitive and psychological outcomes in the awakening and breathing controlled trial. Am J Respir Crit Care Med. 2010 Jul 15;182(2):183-91. doi: 10.1164/rccm.200903-0442OC. Epub 2010 Mar 18. PMID 20299535
- [Background] Schweickert WD, Pohlman MC, Pohlman AS, Nigos C, Pawlik AJ, Esbrook CL, Spears L, Miller M, Franczyk M, Deprizio D, Schmidt GA, Bowman A, Barr R, McCallister KE, Hall JB, Kress JP. Early physical and occupational therapy in mechanically ventilated, critically ill patients: a randomised controlled trial. Lancet. 2009 May 30;373(9678):1874-82. doi: 10.1016/S0140-6736(09)60658-9. Epub 2009 May 14. PMID 19446324
- [Background] Ely EW, Truman B, Shintani A, Thomason JW, Wheeler AP, Gordon S, Francis J, Speroff T, Gautam S, Margolin R, Sessler CN, Dittus RS, Bernard GR. Monitoring sedation status over time in ICU patients: reliability and validity of the Richmond Agitation-Sedation Scale (RASS). JAMA. 2003 Jun 11;289(22):2983-91. doi: 10.1001/jama.289.22.2983. PMID 12799407
- [Background] Vasilevskis EE, Ely EW, Speroff T, Pun BT, Boehm L, Dittus RS. Reducing iatrogenic risks: ICU-acquired delirium and weakness--crossing the quality chasm. Chest. 2010 Nov;138(5):1224-33. doi: 10.1378/chest.10-0466. PMID 21051398
- [Background] Kahn JM, Brake H, Steinberg KP. Intensivist physician staffing and the process of care in academic medical centres. Qual Saf Health Care. 2007 Oct;16(5):329-33. doi: 10.1136/qshc.2007.022376. PMID 17913772
- [Background] Burns KE, Lellouche F, Loisel F, Slutsky AS, Meret A, Smith O, Saskin R, Meade M. Weaning critically ill adults from invasive mechanical ventilation: a national survey. Can J Anaesth. 2009 Aug;56(8):567-76. doi: 10.1007/s12630-009-9124-8. Epub 2009 Jul 7. PMID 19582533
- [Background] Tanios MA, de Wit M, Epstein SK, Devlin JW. Perceived barriers to the use of sedation protocols and daily sedation interruption: a multidisciplinary survey. J Crit Care. 2009 Mar;24(1):66-73. doi: 10.1016/j.jcrc.2008.03.037. Epub 2008 Jun 30. PMID 19272541
- [Background] Mehta S, Burry L, Fischer S, Martinez-Motta JC, Hallett D, Bowman D, Wong C, Meade MO, Stewart TE, Cook DJ; Canadian Critical Care Trials Group. Canadian survey of the use of sedatives, analgesics, and neuromuscular blocking agents in critically ill patients. Crit Care Med. 2006 Feb;34(2):374-80. doi: 10.1097/01.ccm.0000196830.61965.f1. PMID 16424717
- [Background] Thomsen GE, Snow GL, Rodriguez L, Hopkins RO. Patients with respiratory failure increase ambulation after transfer to an intensive care unit where early activity is a priority. Crit Care Med. 2008 Apr;36(4):1119-24. doi: 10.1097/CCM.0b013e318168f986. PMID 18379236
- [Background] Wall RJ, Ely EW, Elasy TA, Dittus RS, Foss J, Wilkerson KS, Speroff T. Using real time process measurements to reduce catheter related bloodstream infections in the intensive care unit. Qual Saf Health Care. 2005 Aug;14(4):295-302. doi: 10.1136/qshc.2004.013516. PMID 16076796
- [Background] Pronovost P, Needham D, Berenholtz S, Sinopoli D, Chu H, Cosgrove S, Sexton B, Hyzy R, Welsh R, Roth G, Bander J, Kepros J, Goeschel C. An intervention to decrease catheter-related bloodstream infections in the ICU. N Engl J Med. 2006 Dec 28;355(26):2725-32. doi: 10.1056/NEJMoa061115. PMID 17192537
- [Background] Barsuk JH, Cohen ER, Feinglass J, McGaghie WC, Wayne DB. Use of simulation-based education to reduce catheter-related bloodstream infections. Arch Intern Med. 2009 Aug 10;169(15):1420-3. doi: 10.1001/archinternmed.2009.215. PMID 19667306
- [Background] Figueroa-Casas JB, Montoya R, Arzabala A, Connery SM. Comparison between automatic tube compensation and continuous positive airway pressure during spontaneous breathing trials. Respir Care. 2010 May;55(5):549-54. PMID 20420724
- [Background] Morris PE, Goad A, Thompson C, Taylor K, Harry B, Passmore L, Ross A, Anderson L, Baker S, Sanchez M, Penley L, Howard A, Dixon L, Leach S, Small R, Hite RD, Haponik E. Early intensive care unit mobility therapy in the treatment of acute respiratory failure. Crit Care Med. 2008 Aug;36(8):2238-43. doi: 10.1097/CCM.0b013e318180b90e. PMID 18596631
- [Background] Strom T, Martinussen T, Toft P. A protocol of no sedation for critically ill patients receiving mechanical ventilation: a randomised trial. Lancet. 2010 Feb 6;375(9713):475-80. doi: 10.1016/S0140-6736(09)62072-9. Epub 2010 Jan 29. PMID 20116842
- [Background] Damschroder LJ, Aron DC, Keith RE, Kirsh SR, Alexander JA, Lowery JC. Fostering implementation of health services research findings into practice: a consolidated framework for advancing implementation science. Implement Sci. 2009 Aug 7;4:50. doi: 10.1186/1748-5908-4-50. PMID 19664226
- [Background] Pun BT, Gordon SM, Peterson JF, Shintani AK, Jackson JC, Foss J, Harding SD, Bernard GR, Dittus RS, Ely EW. Large-scale implementation of sedation and delirium monitoring in the intensive care unit: a report from two medical centers. Crit Care Med. 2005 Jun;33(6):1199-205. doi: 10.1097/01.ccm.0000166867.78320.ac. PMID 15942331
- [Background] Fordis M, King JE, Ballantyne CM, Jones PH, Schneider KH, Spann SJ, Greenberg SB, Greisinger AJ. Comparison of the instructional efficacy of Internet-based CME with live interactive CME workshops: a randomized controlled trial. JAMA. 2005 Sep 7;294(9):1043-51. doi: 10.1001/jama.294.9.1043. PMID 16145024
- [Background] Cook DA, Levinson AJ, Garside S, Dupras DM, Erwin PJ, Montori VM. Internet-based learning in the health professions: a meta-analysis. JAMA. 2008 Sep 10;300(10):1181-96. doi: 10.1001/jama.300.10.1181. PMID 18780847
- [Background] Moore DE Jr, Green JS, Gallis HA. Achieving desired results and improved outcomes: integrating planning and assessment throughout learning activities. J Contin Educ Health Prof. 2009 Winter;29(1):1-15. doi: 10.1002/chp.20001. PMID 19288562
- [Background] Knaus WA, Wagner DP, Draper EA, Zimmerman JE, Bergner M, Bastos PG, Sirio CA, Murphy DJ, Lotring T, Damiano A, et al. The APACHE III prognostic system. Risk prediction of hospital mortality for critically ill hospitalized adults. Chest. 1991 Dec;100(6):1619-36. doi: 10.1378/chest.100.6.1619. PMID 1959406
- [Background] Charlson ME, Pompei P, Ales KL, MacKenzie CR. A new method of classifying prognostic comorbidity in longitudinal studies: development and validation. J Chronic Dis. 1987;40(5):373-83. doi: 10.1016/0021-9681(87)90171-8. PMID 3558716
- [Background] Schoenfeld DA, Bernard GR; ARDS Network. Statistical evaluation of ventilator-free days as an efficacy measure in clinical trials of treatments for acute respiratory distress syndrome. Crit Care Med. 2002 Aug;30(8):1772-7. doi: 10.1097/00003246-200208000-00016. PMID 12163791
- [Background] Harle MT, Dela RF, Veloso G, Rock J, Faulkner J, Cohen MZ. The experiences of Filipino American patients with cancer. Oncol Nurs Forum. 2007 Nov;34(6):1170-5. doi: 10.1188/07.ONF.1170-1175. PMID 18024343
- [Background] Frazier L, Calvin AO, Mudd GT, Cohen MZ. Understanding of genetics among older adults. J Nurs Scholarsh. 2006;38(2):126-32. doi: 10.1111/j.1547-5069.2006.00089.x. PMID 16773915
- [Background] Calvin AO, Frazier L, Cohen MZ. Examining older adults' perceptions of health care providers: identifying important aspects of older adults' relationships with physicians and nurses. J Gerontol Nurs. 2007 May;33(5):6-12. doi: 10.3928/00989134-20070501-03. PMID 17511330
- [Background] Pandharipande PP, Pun BT, Herr DL, Maze M, Girard TD, Miller RR, Shintani AK, Thompson JL, Jackson JC, Deppen SA, Stiles RA, Dittus RS, Bernard GR, Ely EW. Effect of sedation with dexmedetomidine vs lorazepam on acute brain dysfunction in mechanically ventilated patients: the MENDS randomized controlled trial. JAMA. 2007 Dec 12;298(22):2644-53. doi: 10.1001/jama.298.22.2644. PMID 18073360